CLINICAL TRIAL: NCT00668967
Title: Bioequivalence Study Of Verapamil (Covera HS) 240 Mg Extended Release Tablets Produced By Alza Corporation, Vacaville And Pfizer Inc, Puerto Rico: A Two Sequence, Four-Way Crossover Design, Single Dose, Open-Label, Randomized Study In Healthy Volunteers
Brief Title: Bioequivalence Study Of Verapamil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A6661003
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Volunteers
Keywords: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): marketed extended release verapamil tablet
  Interventions: Drug: verapamil
- Test (Other): reformulated extended release verapamil tablet
  Interventions: Drug: verapamil

INTERVENTIONS:
Drug: verapamil — 240 mg extended release tablets once daily at bedtime for 28 days
  Other Names: Covera HS
  Arms: Reference
Drug: verapamil — 240 mg extended release tablets once daily at bedtime for 28 days
  Other Names: Covera HS
  Arms: Test

SUMMARY:
The purpose of this study is to demonstrate bioequivalence of single doses of two verapamil formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* Mass Index (BMI) of approximately 18 to 30 kg/m2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* A positive urine drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Primary study endpoints will be AUClast, AUCinf and Cmax of R- and S-verapamil. | 5 months

SECONDARY OUTCOMES:
Secondary endpoints will include Tmax and t1/2 of R- and S-verapamil and S- and R- norverapamil, as data permit. AUClast, AUCinf and Cmax of R- and S-norverapamil as data permit. | 5 months
Safety and tolerability as assessed by reported adverse events, safety lab test and vital signs | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6661003&StudyName=Bioequivalence%20Study%20Of%20Verapamil